CLINICAL TRIAL: NCT00547820
Title: Urinary Sensor for Cystourethrography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: OBrook2518CTIL
Record Dates: First submitted 2007-10-20; First posted 2007-10-23 (Estimated); Last update posted 2009-10-28 (Estimated); Status verified 2007-10

CONDITIONS: Radiation Dose During VCUG
Keywords: radiation dose; VCUG; pediatric patients

ARMS (2):
- A (Experimental): with application of urinary sensor
  Interventions: Device: Urinary sensor
- B (Placebo Comparator): without use of urinary sensor
  Interventions: Other: placebo

INTERVENTIONS:
Other: placebo
  Arms: B
Device: Urinary sensor
  Arms: A

SUMMARY:
Evaluation of urinary sensor that will be activated by the urine during voiding cystourethrography in pediatric patients

DETAILED DESCRIPTION:
It is of immense importance to perform fluoroscopy during voiding phase of VCUG (Voiding Cystourethrogram) procedures in order to rule out vesicourethral reflux. It is difficult to know exactly when a child will start voiding, so the child is intermittently imaged by fluoroscopy. Fluoroscopy involves radiation, and this we try to diminish as much as possible. We suggest application of small urinary sensor in the perineum of the patient, that will signal the beginning of urination, and only then fluoroscopy will begin. This urinary sensor should cut down substantially radiation dose to the patient.

ELIGIBILITY:
Inclusion Criteria:

* children referred for VCUG procedure at out department

Exclusion Criteria:

* children with pacemakers
* decline to participate

Ages: 1 Month to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2007-07; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Radiation dose during VCUG procedure

CONTACTS AND LOCATIONS:
Overall Officials: Olga R Brook, MD, Principal Investigator — Department of Diagnostic Imaging, Rambam Health Care Campus
Locations (1):
- Department of Diagnostic Imaging, Rambam Health Care Campus, Haifa, Israel